CLINICAL TRIAL: NCT04979416
Title: The Impact of Video Messaging on Vaccination Intention
Brief Title: Video Messages and Vaccination Intention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Mireille Jacobson, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UP-21-00587
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Vaccination

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants do not know if they are in control or treatment or the type of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No video message
- Video message 1 (Experimental)
  Interventions: Behavioral: Video messages
- Video message 2 (Experimental)
  Interventions: Behavioral: Video messages
- Video message 3 (Experimental)
  Interventions: Behavioral: Video messages

INTERVENTIONS:
Behavioral: Video messages — video messages aimed at increasing vaccination
  Arms: Video message 1; Video message 2; Video message 3

SUMMARY:
This study uses an online panel survey to test the impact of video messages on stated likelihood of COVID-19 vaccination. Participants, who have self-identified as unvaccinated against COVID-19, are randomly assigned to either no video message or 1 of 3 video messages to encourage vaccine take-up. The key endpoint is a question about the likelihood of getting vaccinated in the next 30 days.

DETAILED DESCRIPTION:
This study uses an online panel survey to test the impact of video messages on stated likelihood of COVID-19 vaccination. Participants are recruited from the Prolific.co platform. Those who have indicated to Prolific that they have not been vaccinated will be randomly assigned to either no video message or 1 of 3 video messages created by the Vaccinate LA/USC collaborative. The key endpoint is a question about the likelihood of getting vaccinated in the next 30 days.

ELIGIBILITY:
Inclusion Criteria:

* adults in the Prolific.co panel
* unvaccinated against COVID-19

Exclusion Criteria:

* indicated to Prolific.co that they have received a COVID-19 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Vaccination intention | 30 days
  Probability of getting vaccinated in the next 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared after/concurrent with publication.
Supporting Information: Study Protocol, Analytic Code